CLINICAL TRIAL: NCT06408129
Title: COMPArison of Screening Strategies for Active TuBerculosis (COMPASS-TB)
Acronym: COMPASS-TB
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: IRB-MTP_2022_04_202201086
Record Dates: First submitted 2024-04-09; First posted 2024-05-09 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2023-03

CONDITIONS: Active Tuberculosis; Latent Tuberculosis
Keywords: Active Tuberculosis; LAtent Tuberculosis infection; Interferon-Gamma Release Assay; Quantiferon; Chest CT scan; Chest X-ray
MeSH Terms: conditions — Latent Tuberculosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients clinically suspected of active tuberculosis or in contact with index cases: patients had either a clinical suspicion of active tuberculosis or underwent screening due to a close contact with another patient which had a bacteriologically confirmed active tuberculosis.

SUMMARY:
The study is an evaluation of the diagnostic performance of different tests and their association in order to confirm or exclude active tuberculosis.

DETAILED DESCRIPTION:
Background : diagnostic methods to distinguish between latent TB infection (LTBI) and active TB disease remains challenging. Data are scarce concerning the positive predictive value of Current diagnostic approaches, including Interferon-Gamma Release Assay (IGRA) and chest radiography, which is often very low. Computed tomography (CT) scanning, although not recommended by the World Health Organization (WHO) for TB diagnosis, may be of high interest in our high-income low-burden countries. This study assess the performance of the combination of CT scanning and IGRA to diagnose active pulmonary TB and identifies discriminatory CT scan features indicative of active disease.

Methods : A retrospective study was conducted on 580 patients clinically suspected of TB or in contact with bacteriologically confirmed cases (index cases). Patients underwent IGRA testing, thoracic CT scans, and respiratory (or other organs) samples culture. CT scan findings were blindly analyzed, and a composite score combining significant radiological signs with IGRA results was constructed. Diagnostic performance measures, including sensitivity, specificity, positive predictive value (PPV), and negative predictive value (NPV), were calculated.

ELIGIBILITY:
Inclusion Criteria:

Major patients who received the following examinations at the Montpellier University Hospital for tuberculosis screening (clinical suspicion and/or contact with a person with active tuberculosis):

* Chest X-ray AND
* Chest CT scan AND
* Mycobacteriology examination of respiratory or tissue sample (direct/culture/GenXpert) AND
* IGRA test (Quantiferon)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Major patients screened for tuberculosis at the Montpellier University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 580 (Actual)
Dates: Start 2017-01-31 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2024-04-09 (Actual)

PRIMARY OUTCOMES:
Diagnostic performance (sensitivity) of the combination of IGRA and Chest CT scan | Over 12 weeks from the initial medical contact due to suspected tuberculosis to the confirmation or exclusion of this diagnosis
  Sensitivity
Diagnostic performance (specificity) of the combination of IGRA and Chest CT scan | Over 12 weeks from the initial medical contact due to suspected tuberculosis to the confirmation or exclusion of this diagnosis
  specificity

SECONDARY OUTCOMES:
Positive Predictive value of the combination of IGRA and Chest CT scan | Over 12 weeks from the initial medical contact due to suspected tuberculosis to the confirmation or exclusion of this diagnosis
  Positive Predictive value
Negative Predictive value of the combination of IGRA and Chest CT scan | Over 12 weeks from the initial medical contact due to suspected tuberculosis to the confirmation or exclusion of this diagnosis
  Negative Predictive value

CONTACTS AND LOCATIONS:
Overall Officials: Jérémy Charriot, MD, Study Director — University Hospital, Montpellier
Locations (1):
- UH Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: No